CLINICAL TRIAL: NCT06777914
Title: Familial Intrahepatic Cholestasis-related Genes Associated with Disease Susceptibility in Hepato-biliary Cancers
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: HBCs-PFIC; RC-2024-2790618 (Other Grant/Funding Number: Ricerca Corrente 2024 - Ministero della Salute)
Record Dates: First submitted 2024-12-03; First posted 2025-01-16 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2024-11

CONDITIONS: Hepatobiliary Cancers; Progressive Familial Intrahepatic Cholestasis (PFIC); Cholestatic Liver Disease
MeSH Terms: conditions — Cholestasis, progressive familial intrahepatic 1

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — The study involves performing genetic analysis of both the germline, using blood samples, and the somatic, using biopsy material. The biological material for genetic testing will be obtained either through the patient's standard clinical care process or by requesting the patient to provide a study-specific blood sample.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This is a cross-sectional, multicenter tissue study with an exploratory aim to estimate the prevalence of genetic mutations that predispose individuals to diseases in the context of cholestatic disorders and hepatobiliary neoplasms. It is intended as a hypothesis-generating study for future empirical investigations.

DETAILED DESCRIPTION:
This is a multicenter, cross-sectional tissue study designed to explore the prevalence of genetic mutations associated with cholestatic liver diseases and hepatobiliary neoplasms. It aims to generate hypotheses for future empirical research.

Patient data will be collected, including medical history, imaging tests (e.g., abdominal ultrasound, CT, and MRI), and liver function tests, along with [BA] levels. Non-invasive liver fibrosis assessment (FibroScan or Shear-Wave elastography) and, where applicable, liver biopsies will be included, all referenced to the time of genetic testing.

Molecular genetic analysis of PFIC will be conducted using a multiplex PCR NGS panel covering 37 genes. If clinical suspicion remains high despite negative NGS results, Whole Exome Sequencing (WES) will be used to identify previously unknown PFIC-related genes. WES will prioritize patients with hepatobiliary cancers on a healthy liver or without advanced fibrosis and those with a family history of PFIC or related conditions.

Variants will be filtered based on clinical significance, gene-disease associations, and functional predictions, using resources like ClinVar, HGMD, and Personal Genomics PGVD. WES analysis will include at least one affected parent when available, with de novo mutations considered when both parents are involved.

Only pathogenic or potentially pathogenic variants will be reported, confirmed by Sanger sequencing. Genetic counseling will be offered for patients with significant findings. Tumor tissue samples will also be analyzed for somatic mutations, potentially guiding therapeutic decisions or family screening.

NGS for somatic mutations will use tumor samples collected for clinical purposes, with findings compared to germline mutations. This may inform treatment options and surveillance protocols for relatives. The data will be stored in an electronic archive using REDCap and analyzed by clinical staff. The collected data will include clinical history, liver function tests, response to ursodeoxycholic acid, liver fibrosis stage, and molecular results, along with relevant family histories and therapies.

For patients undergoing surgery, the data will also cover pre-operative assessments, surgical techniques, and post-operative outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Instrumental or histological diagnosis of HBCs, defined as primary liver and/or biliary tumors (hepatocellular carcinoma, cholangiocarcinoma, hepatocholangiocarcinoma) occurring in patients without apparent underlying chronic liver disease or in the context of cryptogenic chronic liver disease;
* Curative treatment through surgical resection of the neoplasm or liver transplantation
* Diagnosis of CCLDs defined as:

  1. GGT and/or alkaline phosphatase >1.5 times the normal values in two or more measurements taken at least 6 months apart,
  2. A history of pruritus combined with [BA] >10 mmol/l for a period of ≥6 months.
* Obtaining written informed consent

Exclusion Criteria:

* Other documented causes of chronic liver disease that can justify the clinical phenotype include:

Primary biliary cholangitis Primary sclerosing cholangitis IgG4-related cholangiopathy Obstructive jaundice excluded by the demonstration of normal bile duct anatomy Negative virological tests for HBV, HCV, HEV Alcohol abuse Hemochromatosis Wilson's disease Alpha-1 antitrypsin deficiency

Min Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects with a diagnosis of HBCs who have undergone liver resection or liver transplantation, and a population of patients affected by CCLDs.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2024-10-22 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Pathogenic and Variant Mutations in PFIC Genes in HBCs and CCLDs Patients | 3 years
  To estimate the prevalence of pathogenic germline mutations, probably pathogenic mutations, variants of uncertain significance, probably benign variants, and benign variants in the genes responsible for PFIC in individuals diagnosed with HBCs who have undergone liver resection or liver transplantation, and in a population of patients with CCLDs.

SECONDARY OUTCOMES:
Identifying New PFIC-Associated Genes in HBCs and CCLDs Patients Negative for NGS Analysis via WES | 3 years
  Estimate the percentage of patients carrying newly identified genes potentially responsible for PFIC, discovered through WES
Identification of Somatic Mutations in Tumor Tissue Samples from Patients Undergoing Liver Resection or Transplantation for HBCs | 3 years
  Estimate percentage of patients carrying somatic mutations identified through NGS (in PFIC-related genes) or through WES.
Laboratory and Clinical Features of HBCs and CCLDs Patients | 3 years
  Estimate percentage of patients with PFIC gene mutations and BRIC, LPAC, ICP, DIC phenotype, advanced fibrosis, pruritus, and/or neonatal jaundice
Comparison of Allelic Frequency of PFIC-Related Mutations in the NGS Panel between the Study Population and gnomAD Database | 3 years
  Estimate the proportion of a specific allele among the total alleles identified in the NGS genetic analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Vitale, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (5):
- Italy (5):
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna - Programma Chirurgia addominale nell'insufficienza d'organo terminale e nei pazienti con trapianto d'organo, Bologna, Bologna
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna - UO Chirurgia Epatobiliare e dei Trapianti, Bologna, Bologna
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna - UO Gastroenterologia, Bologna, Bologna
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna - UO Medicina Interna per il trattamento delle gravi insufficienze d'organo, Bologna, Bologna
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna - UO Medicina Interna, malattie epatobiliari e immunoallergologiche, Bologna, Bologna